CLINICAL TRIAL: NCT02346045
Title: Effects of Catheter Based Renal Sympathetic Denervation on Resistant Hypertension in End Stage Renal Disease in Korea
Brief Title: Effect of Renal Denervation in End Staged Renal Disease With Resistant Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry); Daiichi Sankyo Korea Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kiyuk Chang, Professor, chief of division of cardiology, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XC13EIMV0110D; RDN-ESRD-CMC-01 (Other Grant/Funding Number: Daewoong, Daichi-Sankyo)
Record Dates: First submitted 2013-10-21; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Hypertension
Keywords: hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal sympathetic denervation (Experimental): Renal sympathetic denervation procedure plus antihypertensive medication (doses and types of medication are maintained as previously prescribed)
  Interventions: Procedure: Renal sympathetic denervation
- Medical therapy (Sham Comparator): renal angiogram plus antihypertensive medications (doses and types of medication are maintained as previously prescribed)
  Interventions: Procedure: Renal sympathetic denervation

INTERVENTIONS:
Procedure: Renal sympathetic denervation — In the experimental arm, Intervention is renal sympathetic denervation using Symplicity® system (Medtronic Ardian Inc, Mountain View, CA, USA) and antihypertensive medications previously prescribed
  1. After femoral puncture guiding catheter is engaged in renal artery
  2. Symplicity radiofrequency ablation catheter is inserted into renal artery and by circular sequence, from distal to proximal portion, ablation energy is applied to the wall of renal artery
  3. 4-5 ablations are applied in each renal artery.
  In the sham comparator, intervention is renal angiogram and continue antihypertensive medications previuosly decribed
  Other Names: Catheter based based renal sympathetic denervation; Symplicity catheter system by Medtronic

SUMMARY:
A. Hypertension is a major cardiovascular risk factor and numerous treatment strategies have been developed to treat hypertension properly and reduce cardiovascular risk.

B. However, there is a subgroup of hypertension which are resistant to treatment.

1. Resistant hypertension is associated to sympathetic hyperactivity
2. Renal sympathetic nerve is known to be associated with systemic sympathetic activity
3. According to research of recent years, catheter based renal sympathetic denervation is a safe and effective treatment modality to treat resistant hypertension C. Resistant hypertension is observed in end stage renal disease (ESRD) frequently.

D. Sympathetic hyperactivity is observed in ESRD patients E. Catheter based renal sympathetic denervation is expected to improve resistant hypertension in ESRD patients

F. The aim the present study is to evaluate the effects and safety of catheter based renal sympathetic denervation on resistant hypertension in ESRD

ELIGIBILITY:
Inclusion Criteria:

* Patients who are under hemodialysis due to end stage renal disease
* Patients who have resistant hypertension with office SBP >160 mmHg)
* Patients who are or over 18 years old.
* Patients who submit informed consent

Exclusion Criteria:

* Known secondary hypertension patients
* Patients who have renal artery which is not adequate for renal denervation

  1. The main renal artery diameter < 4 mm, or renal artery length < 20 mm
  2. The renal arteries into which stable catheter insertion is difficulty and which have hemodynamically or anatomically significant stenosis
  3. The renal arteries who have undergone renal angioplasty
* Patients who have history of myocardial infarction, unstable angina, syncope cerebrovascular insufficiency or extensive atherosclerotic disease with intravascular thrombosis, or unstable plaque
* Type 1 Diabetes
* Patients who have scheduled percutaneous coronary intervention (PCI) or operation within 6 months
* Hemodynamically significant valvular heart disease in which blood pressure reduction may cause significant deterioration of patient's health.
* Primary pulmonary hypertension
* Patients who have the intracardiac defibrillator(ICD) or pacemaker which do not allow delivery of radiofrequency energy.
* Patients who require continuous oxygen supply or mechanical ventilation for treatment of obstructive sleep apnea
* Patients who have serious medical condition which can compromise the safety of the patients and the safety and integrity of the study.
* Patients who have unresolved drug issue, alcoholism
* Patients who lack ability to understand and follow the instruction the researcher
* Patient who cannot follow up
* Patients who are registered in other trial
* Patients who are pregnant, nursing or planning to be pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-08 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
The change of office systolic blood pressure after renal denervation | 6 month

SECONDARY OUTCOMES:
Change of office diastolic blood pressure | 6 month
change in ambulatory blood pressure monitroing(ABPM): mean systolic blood pressure(SBP)/diastolic blood pressure(DBP), mean heart rate(HR), BP variability | 6 month
Change in plasma norepinephrine | 6 months
Change in pulse wave velocity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiyuk Chang, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital; Sung Ho Her, MD, PhD, Principal Investigator — Daejon St. Mary's Hospital
Locations (4):
- South Korea (4):
  - Daejon St. Mary's Hospital, Daejeon, Chungchung Nam Do
  - Chungnam National University, Daejeon, Chungchungnamdo
  - Pohang St. Mary's Hospital, Pohang, Kyungsangnamdo
  - Seoul St. Mary's Hospital, Seoul, Seoul

REFERENCES:
- [Background] Schlaich MP, Bart B, Hering D, Walton A, Marusic P, Mahfoud F, Bohm M, Lambert EA, Krum H, Sobotka PA, Schmieder RE, Ika-Sari C, Eikelis N, Straznicky N, Lambert GW, Esler MD. Feasibility of catheter-based renal nerve ablation and effects on sympathetic nerve activity and blood pressure in patients with end-stage renal disease. Int J Cardiol. 2013 Oct 3;168(3):2214-20. doi: 10.1016/j.ijcard.2013.01.218. Epub 2013 Feb 28. PMID 23453868
- [Background] Esler MD, Krum H, Schlaich M, Schmieder RE, Bohm M, Sobotka PA; Symplicity HTN-2 Investigators. Renal sympathetic denervation for treatment of drug-resistant hypertension: one-year results from the Symplicity HTN-2 randomized, controlled trial. Circulation. 2012 Dec 18;126(25):2976-82. doi: 10.1161/CIRCULATIONAHA.112.130880. PMID 23248063
- [Background] Symplicity HTN-1 Investigators. Catheter-based renal sympathetic denervation for resistant hypertension: durability of blood pressure reduction out to 24 months. Hypertension. 2011 May;57(5):911-7. doi: 10.1161/HYPERTENSIONAHA.110.163014. Epub 2011 Mar 14. PMID 21403086